CLINICAL TRIAL: NCT00465283
Title: Donepezil Double Blind Trial for ECT Memory Disfunction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: BeerYaakov Mental Health Center (Other Government)
Responsible Party: Marina Kupchik, MD, BeerYaakov Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Donepezil-180CTIL
Record Dates: First submitted 2007-04-22; First posted 2007-04-24 (Estimated); Last update posted 2009-01-27 (Estimated); Status verified 2009-01

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder
Keywords: Donepezil, ECT, Memory Disfunction
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Epilepsy, Rolandic | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Donepezil (Active Comparator)
  Interventions: Drug: Donepezil
- placebo (Placebo Comparator)
  Interventions: Drug: Donepezil

INTERVENTIONS:
Drug: Donepezil — Tab.Donepezil 5 mg once daily during ECT treatment and the month after the last ECT treatment
  Other Names: Donepezil - Memorit

SUMMARY:
This is a double blind randomized investigation of donepezil for patients suffering from schizophrenia, undergoing ECT.

Patients will be randomized to receive either donezepil or plasebo, in order to gauge whether donezepil has a protective effect on memory disfunction, while patients are treated with ECT. Several parameters will be invistigated at baseline: general psychopathological measures, memory function scales, side effects scales. The same measurements will be taken throughout the trial and one month after ending the ECT.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia, Schizoaffective disorder, schizophreniform disorder patients who meet criteria for diagnoses by DSM-IV criteria and evaluated by the Structured Clinical Interview for DSM-IV (SCID)

Exclusion Criteria:

* History of serious neurological disorders including neurodegenerative deseases, mental retardation, substance and/or alcohol dependence.
* Pregnant women
* Patients who recieved ECT within 6 month
* Patients whith contraindication to Donepezil treatment.
* Patients with Lithium treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-05; Primary Completion 2010-01 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Data will be analyzed using SPSS for Windows. | after 5 ECT treatments
Results of the memory and neurocognitive measures will be examined | after 8 ECT treatments
using repeated MANOVA with before, within and after ECT treatment. | 1 month after the last ECT treatment

CONTACTS AND LOCATIONS:
Overall Officials: Tali Nachshoni, MD, Principal Investigator — Beer Yaakov Mental Health Center
Locations (1):
- Beer Yaakov MHC, Beer Yaacov, Israel